CLINICAL TRIAL: NCT07048769
Title: Paracervical Block for Saline Infusion Sonogram in Fertility Evaluation: A Randomized Controlled Trial
Brief Title: Paracervical Block for Pain Reduction in Saline Infusion Sonograms
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024-16284
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Pain During Saline Infusion Sonogram
Keywords: paracervical block; saline infusion sonogram; Fertility evaluation
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: Participants are randomized in a 1:1 ratio to receive either a lidocaine paracervical block or no anesthesia during saline infusion sonogram. Each participant receives only one intervention.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Paracervical Block Arm (Experimental): Participants receive a paracervical block with 10cc 1% lidocaine buffered with 1cc sodium bicarbonate
  Interventions: Drug: Lidocaine
- Control Arm (No Block) (Placebo Comparator): Participants receive no anesthesia; a capped needle is pressed at the paracervical locations to mimic injection
  Interventions: Procedure: Sham paracervical block

INTERVENTIONS:
Drug: Lidocaine — 10cc of 1% lidocaine buffered with 1cc 8.4% sodium bicarbonate, injected at 4 and 8 o'clock paracervical positions.
  Arms: Paracervical Block Arm
Procedure: Sham paracervical block — A capped needle is pressed at 4 and 8 o'clock positions to mimic lidocaine block without injection.
  Arms: Control Arm (No Block)

SUMMARY:
Inadequate pain management during gynecologic procedures is a growing women's health concern, especially as it reduces access to care for patients who may subsequently avoid further treatment. Although recent evidence has shown that local anesthesia reduces pain during certain gynecologic procedures, such as intrauterine (IUD) placements, there is still limited evidence on the effectiveness of local anesthesia during saline infusion sonograms (SIS). The SIS is a routine procedure performed during the fertility workup to evaluate the uterus and fallopian tubes. In this study, the investigators are determining if local anesthesia improves the pain experience for women undergoing SIS by randomly assigning 246 women to receive local anesthesia (lidocaine) versus placebo (capped needle pressing against areas where the paracervical block is performed). The investigators will compare their self-reported pain scores at various points in the procedure. If local anesthesia is shown to be effective at reducing pain, this could ultimately improve the patient experience in fertility evaluations moving forward and make this procedure more accessible to all women.

DETAILED DESCRIPTION:
Pain management options (or lack thereof) during routine gynecologic procedures has become a women's health concern with growing prominence. Patients increasingly are reporting their "excruciating" pain experiences from gynecologic procedures ranging from pap smears to intrauterine device placements. When pain during gynecologic procedures is not well managed, gynecologic care quality and frequency suffers - one study found that in a group of middle-aged black women, those who perceived pap smears to be painful were almost five times more likely to not adhere to regular pap screening recommendations. Women, similarly, may avoid other elective gynecologic procedures, such as intrauterine device placement or saline infusion sonograms, out of fear of pain during the procedure.

Recent evidence has found that local anesthesia can significantly reduce pain during certain procedures, such as surgical abortion and intrauterine device placement (IUD). For example, in two randomized controlled trials of nulliparous women undergoing intrauterine device placement, a 10-20cc buffered 1% lidocaine paracervical block decreased pain during and following IUD placement. However, this reduction in pain may not be significant in multiparous women-in systematic review and meta-analysis of randomized clinical trials (RCTs) of pain management options for women undergoing IUD placement, paracervical blocks were not found to reduce pain in a statistically significant fashion. In women undergoing surgical abortion, a 20cc 1% lidocaine injection significantly reduced pain during dilation and aspiration regardless of parity status.

In reproductive endocrinology and infertility offices, saline infusion sonogram is often performed in the evaluation of uterine cavity and patency of the fallopian tubes. This is a procedure that is demonstrated to cause mild to moderate pain in most patients. These procedures do not standardly receive any local anesthesia, though many practices will recommend an over-the-counter nonsteroidal anti-inflammatory drug (NSAID) prior to procedure. Although no previous study has been published on NSAIDs specifically, a prospective observational study did find that pre-medication of paracetamol + codeine prior to saline ultrasound assessment of uterine cavity and tubal patency significantly reduced pain.

While local anesthesia is not routinely offered during these saline infusion sonograms, several studies have investigated its potential effect. One randomized controlled trial assessed the pain relief effect of topical and intrauterine lidocaine during saline ultrasound, and found no difference in pain compared to placebo. Of note, these saline ultrasounds were only for cavity evaluation, not tubal evaluation, and therefore did not utilize a balloon catheter. Another randomized controlled trial of 96 Turkish women found that paracervical block significantly reduced pain during saline infusion sonogram compared to the placebo group. However, of note, this protocol utilized a tenaculum, which is not routinely used in saline infusion sonograms in the United States for fertility evaluation. Additionally, the catheter diameter used was wider than is used in the clinic (4mm versus 1.67mm). This study also did not appear to evaluate for tubal patency, as the catheter described was not a balloon catheter.

In this study, the investigators aim to add to the existing literature on pain management during saline infusion sonograms to determine if lidocaine paracervical blocks decrease perceived pain in saline ultrasounds that assess for uterine cavity and tubal patency. This will be accomplished by determining if paracervical block provides clinically significant pain relief compared to no anesthesia during saline ultrasound evaluation of uterine cavity and tubal patency.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing uterine cavity and tubal patency evaluation via saline infusion sonogram with balloon catheter at Montefiore Institute for Reproductive Medicine and Health
* Pre-medicated with 600-800 mg ibuprofen taken 30 minutes to 4 hours prior to procedure
* Able to provide informed consent in English or Spanish
* Capacity to consent

Exclusion Criteria:

* Undergoing uterine cavity evaluation only (without tubal patency assessment)
* No ibuprofen pre-medication prior to procedure
* Received misoprostol within 24 hours prior to procedure
* Known allergy to lidocaine

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 246 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity from baseline during tubal patency assessment | Measured during the procedure, within 30 minutes of procedure start
  Pain intensity during tubal patency assessment will be assessed using a Visual Analog Scale (VAS) ranging from 0 to 100 mm, where 0 represents "no pain" and 100 represents "worst possible pain." The VAS score will be recorded at the time of saline infusion sonogram assessing tubal patency. The pain intensity will be evaluated as a change from their baseline level of pain. Results will be summarized by study arm and analyzed using basic descriptive statistics.

SECONDARY OUTCOMES:
Pain intensity during paracervical block administration | This will be obtained during the procedure, usually within 10 minutes of procedure start.
  Pain intensity during paracervical block administration will be assessed using a Visual Analog Scale (VAS) ranging from 0 to 100 mm, where 0 represents "no pain" and 100 represents "worst possible pain." The VAS score will be measured at the time of paracervical block injection or needle pressure. Results will be summarized by study arm and analyzed using basic descriptive statistics.
Pain intensity during balloon catheter placement | This will be obtained during the procedure, typically within 10 minutes of procedure start
  Pain intensity during balloon catheter placement will be assessed using a Visual Analog Scale (VAS) ranging from 0 to 100 mm, where 0 represents "no pain" and 100 represents "worst possible pain." The VAS score will be recorded at the time of balloon catheter placement. Results will be summarized by study arm and analyzed using basic descriptive statistics.
Pain intensity during saline infusion for uterine cavity assessment | This will be obtained during the procedure, within 30 minutes of procedure start
  Pain intensity during saline infusion for uterine cavity assessment will be assessed using a Visual Analog Scale (VAS) ranging from 0 to 100 mm, where 0 represents "no pain" and 100 represents "worst possible pain." The VAS score will be recorded at the time of uterine cavity assessment. Results will be summarized by study arm and analyzed using basic descriptive statistics.
Pain intensity upon completion of the procedure | This will be obtained during the procedure, typically within 30 minutes of procedure start
  Pain intensity will be assessed using a Visual Analog Scale (VAS) ranging from 0 to 100 mm, where 0 represents "no pain" and 100 represents "worst possible pain." The VAS score will be recorded at procedure completion. Results will be summarized by study arm and analyzed using basic descriptive statistics.
Pain intensity 1 hour after procedure | Approximately 1 hour following the procedure
  Pain intensity following the procedure will be assessed using a Visual Analog Scale (VAS) ranging from 0 to 100 mm, where 0 represents "no pain" and 100 represents "worst possible pain." The VAS score will be recorded 1 hour after procedure completion. Results will be summarized by study arm and analyzed using basic descriptive statistics.
Percentage of patients not able to receive the paracervical block | This will be determined on day of procedure, typically within 10 minutes of procedure start
  Paracervical blocks sometimes cannot be completed due to anatomic challenges If patients in the lidocaine intervention group are not able to receive the paracervical block due to anatomical challenges, this will be recorded. The percentage of patients who are not able to receive the paracervical block will be summarized using basic descriptive statistics.
Percentage of patients requiring tenaculum for catheter insertion | This will be obtained during the procedure, typically within 10 minutes of procedure start
  Some patients require tenaculum (a metal two-prong grasper) placement on the cervix in order the for the balloon catheter of the saline infusion sonogram to be inserted into the uterine cavity. Whether a tenaculum was used will be recorded. The percentage of participants for whom tenaculum was used to facilitate catheter placement will be summarized using basic descriptive statistics.
Percentage of patients for whom uterine sound was used to complete the saline ultrasound | This will be collected during the procedure, within 30 minutes of procedure start
  Some patients for whom there is initial difficulty in entering the uterine cavity with a balloon catheter require use of a uterine sound to map the cervical canal prior to placing the balloon catheter. The percentage of patients for whom a uterine sound is used will be recorded and analyzed using basic descriptive statistics.

OTHER OUTCOMES:
Patient satisfaction with pain control method | Within 1 hour of procedure completion
  Patients will complete a survey within 1 hour of procedure completion asking if they would choose the same pain control method again, with options of "yes", "no" and "unsure". Responses will be summarized and analyzed using basic descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Julian Gingold, MD, PhD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore's Institute for Reproductive Medicine and Health, Hartsdale, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
Decisions about IPD sharing will be made after the study's completion. Updates regarding data sharing plans will be provided as they become available.

REFERENCES:
- [Background] Ozkan S, Kars B, Sakin O, Onan Yilmaz A, Bektas YT, Kasikci HO. The optimal analgesic method in saline infusion sonogram: A comparison of two effective techniques with placebo. Turk J Obstet Gynecol. 2016 Sep;13(3):132-136. doi: 10.4274/tjod.46667. Epub 2016 Sep 15. PMID 28913108
- [Background] Yung SS, Lai SF, Lam MT, Lee VC, Li RH, Ho PC, Ng EH. Randomized, controlled, double-blind trial of topical lidocaine gel and intrauterine lidocaine infusion for pain relief during saline contrast sonohysterography. Ultrasound Obstet Gynecol. 2016 Jan;47(1):17-21. doi: 10.1002/uog.15775. Epub 2015 Nov 29. PMID 26434382
- [Background] Ludwin I, Martins WP, Nastri CO, Ludwin A. Pain Intensity During Ultrasound Assessment of Uterine Cavity and Tubal Patency With and Without Painkillers: Prospective Observational Study. J Minim Invasive Gynecol. 2017 May-Jun;24(4):599-608. doi: 10.1016/j.jmig.2017.01.015. Epub 2017 Feb 1. PMID 28159714
- [Background] Rogerson L, Bates J, Weston M, Duffy S. A comparison of outpatient hysteroscopy with saline infusion hysterosonography. BJOG. 2002 Jul;109(7):800-4. doi: 10.1111/j.1471-0528.2002.01478.x. PMID 12135217
- [Background] Renner RM, Nichols MD, Jensen JT, Li H, Edelman AB. Paracervical block for pain control in first-trimester surgical abortion: a randomized controlled trial. Obstet Gynecol. 2012 May;119(5):1030-7. doi: 10.1097/AOG.0b013e318250b13e. PMID 22525915
- [Background] Samy A, Abbas AM, Mahmoud M, Taher A, Awad MH, El Husseiny T, Hussein M, Ramadan M, Shalaby MA, El Sharkawy M, Hatem D, Alaa-El-Din Wali A, Abd-El-Fatah SM, Hussein AH, Haggag H. Evaluating different pain lowering medications during intrauterine device insertion: a systematic review and network meta-analysis. Fertil Steril. 2019 Mar;111(3):553-561.e4. doi: 10.1016/j.fertnstert.2018.11.012. Epub 2019 Jan 2. PMID 30611553
- [Background] Akers AY, Steinway C, Sonalkar S, Perriera LK, Schreiber C, Harding J, Garcia-Espana JF. Reducing Pain During Intrauterine Device Insertion: A Randomized Controlled Trial in Adolescents and Young Women. Obstet Gynecol. 2017 Oct;130(4):795-802. doi: 10.1097/AOG.0000000000002242. PMID 28885425
- [Background] Mody SK, Farala JP, Jimenez B, Nishikawa M, Ngo LL. Paracervical Block for Intrauterine Device Placement Among Nulliparous Women: A Randomized Controlled Trial. Obstet Gynecol. 2018 Sep;132(3):575-582. doi: 10.1097/AOG.0000000000002790. PMID 30095776
- [Background] Hoyo C, Yarnall KS, Skinner CS, Moorman PG, Sellers D, Reid L. Pain predicts non-adherence to pap smear screening among middle-aged African American women. Prev Med. 2005 Aug;41(2):439-45. doi: 10.1016/j.ypmed.2004.11.021. PMID 15917039
- [Background] O'Donohue S. The ripples of trauma caused by severe pain during IUD procedures. BMJ. 2021 Aug 5;374:n1910. doi: 10.1136/bmj.n1910. No abstract available. PMID 34353791
- [Background] Nudson, Rae. Gynecology Has a Pain Problem. The Cut, Jun 1 2022.